CLINICAL TRIAL: NCT02170454
Title: Effect of Pharyngeal Cortical Area Inhibition Induced by rTMS on Swallowing Function in Healthy Subject: Video Fluoroscopic Study.
Brief Title: Effect of Pharyngeal Inhibition by rTMS on Swallowing Function
Acronym: rTMSvideoSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2007/055/HP
Record Dates: First submitted 2009-02-17; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Oropharyngeal Dysphagia
Keywords: neuromodulation; swallowing; magnetic stimulation; healthy subjects
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS (Active Comparator): rTMS on pharyngeal cortical area in healthy subjects
  Interventions: Procedure: magnetic stimulation
- Placebo (Placebo Comparator): Sham rTMS on pharyngeal cortical area in healthy subjects
  Interventions: Procedure: magnetic stimulation

INTERVENTIONS:
Procedure: magnetic stimulation — rTMS on pharyngeal cortical area in healthy subjects or sham rTMS on pharyngeal cortical area in healthy subjects

SUMMARY:
The aim of this study is to test the hypothesis that rTMS on the dominant swallowing hemisphere is able to modify swallowing coordination.

DETAILED DESCRIPTION:
The aim of the study is to demonstrate that rTMS (on the dominant hemisphere, on the nondominant hemisphere and placebo rTMS) are able to modify swallowing coordination on healthy subjects. Swallowing function will be studied before and after rTMS with videomanometry.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* healthy subjects

Exclusion Criteria:

* epilepsia
* brain injury
* stroke
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
pharyngeal pressure | Day 1
  Swallowing function will be studied before and after rTMS with videomanometry

SECONDARY OUTCOMES:
swallowing time | Day 1
  Swallowing function will be studied before and after rTMS with videomanometry

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, MDPhD, Principal Investigator — Rouen University
Locations (1):
- VERIN, Rouen, France